CLINICAL TRIAL: NCT04268277
Title: Pembrolizumab in Marginalzone Lymphoma a MULTICENTER OPEN LABEL SINGLE-ARM PHASE II STUDY
Brief Title: Pembrolizumab in MarginalzoneLymphoma a MULTICENTER OPEN LABEL SINGLE-ARM PHASE II STUDY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to slow recruitment caused by the COVID-19 pandemic and associated retrictions and the authorization of zanubrutinib. Additionally, many competing trials promising higher efficacy have been started in the meantime.
Sponsor: University of Ulm (Other)
Collaborators: X-act Cologne Clinical Research GmbH (Industry); Zentrum für Klinische Studien Ulm (Other); Merck Sharp & Dohme LLC (Industry); Celltrion Healthcare Co., LTD (Unknown)
Responsible Party: Principal Investigator, Christian Buske, Prof. Dr., University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLE-1
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Marginal Zone Lymphoma
Keywords: Hematology; Oncology; Relapse; MALT; Pembrolizumab; Rituximab
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Neoplasms; Recurrence | interventions — Rituximab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rituximab & Pembrolizumab (Experimental): Cycle 1 (21 days cycle):
  Rituximab: 375 mg/m2 day 1, 8, 15 Pembrolizumab: 200 mg IV fixed dose day 2
  Cycle 2-18 (21 days cycle) or until progression or non-tolerable toxicity:
  Rituximab: 375 mg/m2 day 1 every second cycle Pembrolizumab: 200 mg IV fixed dose day 1
  Interventions: Drug: Rituximab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Rituximab — 100 mg concentrate for solution for infusion
  Other Names: Truxima
Drug: Pembrolizumab — 100 mg/ 4mL concentrate for solution for infusion
  Other Names: Keytruda

SUMMARY:
For marginal zone lymphoma (MZL) Rituximab in combination with conventional chemotherapy is widely used for those patients who fail local therapy or do not qualify for such. Depending on the MZL subtype Rituximab/chemotherapy is able to induce in part long remissions, but does not prevent relapse later on. In addition, chemotherapy associated toxicity is often problematic in MZL patients, who are mostly of advanced age. Thus, chemotherapy-free approaches are highly attractive for this patient group. Rituximab single agent is a widely used chemotherapy-free approach in MZL, but was significantly inferior compared to Rituximab/chlorambucil in a large randomized prospective clinical trial in treatment naïve MZL with a CR rate of 55.8% vs. 78.8%, respectively (P < 0.001). Thus, it is the major aim to develop chemotherapy-free approaches for MZL, which approach or surpass efficacy of rituximab/chemotherapy combinations, but avoid chemotherapy associated toxicities.

Checkpoint inhibitors such as Pembrolizumab have revolutionized cancer treatment and have also shown first encouraging results in Non-Hodgkin lymphomas. Based on these observations it is the aim of this study to test the toxicity and efficacy of Pembrolizumab in combination with the anti-CD20 antibody Rituximab in patients with newly diagnosed or relapsed MZL in need of treatment, who are not eligible or failed local therapy, following the assumption that this novel chemotherapy-free combination is significantly more efficient than Rituximab single agent therapy and at least as efficient as rituximab/chemotherapy, but avoids chemotherapy-related toxicity.

DETAILED DESCRIPTION:
For marginal zone lymphoma (MZL) Rituximab in combination with conventional chemotherapy is widely used for those patients who fail local therapy or do not qualify for such. Depending on the MZL subtype Rituximab/chemotherapy is able to induce in part long remissions, but does not prevent relapse later on. In addition, chemotherapy associated toxicity is often problematic in MZL patients, who are mostly of advanced age. Thus, chemotherapy-free approaches are highly attractive for this patient group. Rituximab single agent is a widely used chemotherapy-free approach in MZL, but was significantly inferior compared to Rituximab/chlorambucil in a large randomized prospective clinical trial in treatment naïve MZL with a CR rate of 55.8% vs. 78.8%, respectively (P < 0.001). Thus, it is the major aim to develop chemotherapy-free approaches for MZL, which approach or surpass efficacy of rituximab/chemotherapy combinations, but avoid chemotherapy associated toxicities.

Checkpoint inhibitors such as Pembrolizumab have revolutionized cancer treatment and have also shown first encouraging results in Non-Hodgkin lymphomas. Based on these observations it is the aim of this study to test the toxicity and efficacy of Pembrolizumab in combination with the anti-CD20 antibody Rituximab in patients with newly diagnosed or relapsed MZL in need of treatment, who are not eligible or failed local therapy, following the assumption that this novel chemotherapy-free combination is significantly more efficient than Rituximab single agent therapy and at least as efficient as rituximab/chemotherapy, but avoids chemotherapy-related toxicity.

The objective of the trial is to test the efficacy and toxicity of treatment with Pembrolizumab and Rituximab in patients with MZL in need of treatment, who have failed or are not eligible for local therapy or relapsed. For efficacy the rate of complete remissions (according to the GELA criteria for gastric MALT or to the Cheson 2007 criteria for nodal and splenic MZL) after end of treatment (18 cycles) will be primarily analyzed. For toxicity assessment treatment associated adverse events, quality of life and cumulative incidence of secondary malignancies will be documented.

This study is a European multicenter, single-arm, open-label, phase II trial of 18 cycles of Pembrolizumab and Rituximab in patients aged ≥ 18 years with previously untreated or relapsed MZL in need of treatment.

Primary endpoint is the complete response (CR rate (CRR) determined after end of treatment (18 cycles).

The study flow will be as follows:

* Previously untreated or relapsed patients will be screened for eligibility for the trial. If the patient is eligible for the study, the patient will be registered before the first cycle of treatment.
* Patients who progress at any time point during treatment are considered as treatment failure. They will be followed up for overall survival until end of follow up period or death.
* Patients, who achieve at least a SD after treatment will be followed up for response until progression/relapse and for overall survival until death.

It is expected that a total of 56 patients at approximately 15 investigator sites in Germany and 3 centers in Austria will be registered. Every patient will receive treatment over a time period of 18 cycles (each cycle lasts 3 weeks). Subsequently, patients will be monitored every 3 months for 2 additional years, subsequently every 6 months for three additional years. The follow-up phase will be shorter than 5 years if End of Study is reached before this time period.

ELIGIBILITY:
Inclusion Criteria:

Patients must have a proven pathological diagnosis of MZL, diagnosed by a reference pathology center.

Patients must meet the following inclusion criteria to be eligible for participation in this study:

* Confirmed CD20 positive de novo or relapsed MALT Lymphoma in need of treatment following or being not eligible for local therapy (including surgery, radiotherapy and antibiotics e.g. for H. pylori-positive gastric lymphoma arisen at any extranodal site) OR
* Confirmed CD20 positive de novo or relapsed splenic MZL in need of treatment following or not being eligible for local therapy (including surgery and antiviral therapy for Hepatitis C Virus) OR
* Confirmed CD20 positive de novo or relapsed nodal MZL in need of treatment following or not being eligible for local therapy (radiotherapy). The need of treatment is applicable in the case of B symptoms, deterioration of peripheral blood counts due to lymphoma infiltration of the bone marrow, rapid enlargement of lymph nodes or compression of vital organs by bulky disease.

For nodal MZL and extragastric MALT lymphoma:

• At least one bi-dimensionally measurable lesion (>=1.5 cm in its largest dimension by CT/PET-CT scan or MRI)

For splenic MZL (SMZL):

In patients with splenic MZL, an enlarged spleen on CT scan and lymphoma cell infiltration has to be seen in bone marrow and/or peripheral blood.

At least one of the following criteria must be fulfilled:

* Bulky progressive or painful splenomegaly
* one of the following symptomatic/progressive cytopenias: Hb < 10 g/dL, or Platelet count < 80.000 /µL, or neutropenia < 1000 /µL, whatever the reason (autoimmune or hypersplenism or bone marrow infiltration)
* splenectomised patients with rapidly raising lymphocyte counts, development of lymphadenopathy or involvement of extranodal sites if not being eligible for local therapy
* SMZL with concomitant hepatitis C infection which has not responded to or has relapsed after Interferon and/or Ribavirin and/or direct antiviral agents (patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA)

For gastric MALT Lymphoma:

For gastric MALT lymphoma, the clinical evidence of the MZL as seen by gastroendoscopy is sufficient. There is no need to show a measurable lesion by CT scan or MRI.

Inclusion is possible for patients with:

* H. pylori-negative cases following or being not eligible for local therapy (i.e., surgery, radiotherapy or antibiotics) or after systemic therapy
* H. pylori-positive disease that has remained stable, progressed, or relapsed following antibiotic therapy

Others:

* Age ≥ 18 years
* Life expectancy > 3 months
* Meet the following pretreatment laboratory criteria at the Screening visit conducted within 28 days of study enrollment (unless due to underlying lymphoma):

  * Baseline platelet count ≥ 75 x 109/L (if not due to BM infiltration by the lymphoma), absolute neutrophil count ≥ 1.5 x 109/L.
  * Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L (Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks)
  * International Normalized Ratio (INR) or Prothrombin Time (PT): ≤ 1.5 × ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT): ≤ 1.5 × ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * ASAT (SGOT): ≤ 2.5 times the upper limit of institutional laboratory normal value or ≤ 5 times the upper limit of institutional laboratory normal value in subjects with lymphoma in the liver.
  * ALAT (SGPT): ≤ 2,5 times the upper limit of institutional laboratory normal value or ≤ 5 times the upper limit of institutional laboratory normal value in subjects with lymphoma in the liver
  * Serum total bilirubin: ≤ 1.5 × ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN (unless clearly related to the disease)
  * Serum creatinine ≤ 1.5 × ULN OR ≥ 60 mL/min GFR or CrCl for subjects with creatinine levels > 1.5 × institutional ULN
  * Negative HIV antibody
  * Patients with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) may be included if HBV DNA is undetectable, provided that they are willing to undergo monthly DNA testing. Patients who have protective titers of HBSAb after vaccination or prior but cured hepatitis B are eligible.
  * Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
  * For women of child-bearing potential only: Pregnancy β-HCG negative. Serum or urine β-HCG must be negative during screening and at study enrolment visit.
* Premenopausal fertile females must agree to use a highly effective method of birth control for the duration of the therapy up to 12 months after the last dose of Rituximab and through 4 months after the last dose of Pembrolizumab. A highly effective method of birth control is defined as those which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomised partner or sexual abstinence. Contraception and pregnancy testing are required according the CTFG recommendations (http://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf)
* Men must agree not to father a child for the duration of therapy and 6 months after and must agree to advice a female partner to use a highly effective method of birth control. According to CTFG recommendations, men must use condoms.
* Willingness and ability to comply with scheduled visits, drug administration plan, imaging studies, laboratory tests, other study procedures, and study restrictions
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential benefits, possible side effects, potential risks and discomforts, and other pertinent aspects of study participation

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrolment:

* ECOG performance status ≥ 2
* History of a malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate specific antigen for ≥ 1 year prior to study enrolment visit, other malignancy treated with a curative intent and currently in complete remission, for ≥ 3 years
* Central nervous system lymphoma, leptomeningeal lymphoma, or histologic evidence of transformation to a high-grade or diffuse large B-cell lymphoma
* Has had prior chemotherapy (systemic anti-cancer therapy), targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or baseline value) from AEs due to a previously administered agent

  * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If a subject received major surgery, they must have recovered adequately from complications from the intervention prior to starting therapy
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of study enrolment visit
* Ongoing drug-induced liver injury, chronic active hepatitis B (HBV), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cholangitis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension
* Treatment with any other investigational agent or participating in another clinical trial with an investigational product within 4 weeks prior to entering this study or within 5 x the half-life (t1/2) of the investigational product, whichever is longer
* Breastfeeding or Pregnancy
* Congestive heart failure > New York Heart Association (NYHA) class 2
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months)
* Myocardial infarction less than 6 months before start of study medication
* Uncontrolled arterial hypertension despite optimal medical management
* Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, electrocardiogram (ECG) finding, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the subject or impair the assessment of study results
* Vaccination with a live vaccine within 30 days prior to start of therapy
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication
* Non-healing wound, ulcer, or bone fracture
* History or concurrent interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator)
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137)
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment
* Has a history of non-infectious pneumonitis that required steroids, or current pneumonitis
* History of anaphylaxis in association with previous administration of monoclonal antibodies or severe hypersensitivity (≥Grade 3) to the investigational medicinal products and/or any of its excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a known history of active TB (Bacillus Tuberculosis)
* Medical history of allogeneic stem cell transplant
* Ongoing alcohol or drug addiction or known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Diagnosis of Stevens-Johnson Syndrome (SJS) and Toxic Epidermal Necrolysis (TEN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
CR rate | 12 months
  CR rate (CRR) after end of treatment (18 cycles)

SECONDARY OUTCOMES:
Response rate | 58 weeks
  The response rates are evaluated 4 weeks after the end of treatment
Best response | 54 weeks
  Best response is determined in the time interval from the start of induction therapy to end of follow-up.
Time to best response | 54 weeks
  Time to best response is defined as the time from the start of induction to best response the patient achieves (CR, PR)
Time to first response | 54 weeks
  Time to first response is defined as the time from the start of induction to first response (CR, PR)
Progression free survival (PFS) | 54 weeks
  Progression free survival (PFS) is defined as the time from registration to the first occurrence of progression or relapse as assessed by the investigator, or death from any cause. PFS for patients without disease progression, relapse, or death will be censored at the time of the last tumor assessment.
Time to treatment failure (TTF) | 54 weeks
  Time to treatment failure is defined as the time of registration to discontinuation of therapy for any reason including death from any cause, progression, toxicity or add-on of new anti-cancer therapy. Patients alive without treatment failure are censored at the latest tumor assessment date.
Duration of Response (DR) | 54 weeks
  Duration of response will be calculated in patients with response (CR, PR) to induction from end of induction to the date of progression, relapse or death from any cause. Patients alive without progression and relapse will be censored at the latest tumor assessment date or the stopping date.
Cause specific survival (CSS) | 54 weeks
  Cause specific survivial is defined as the period from the induction registration to death from lymphoma or lymphoma related cause; death unrelated to MZL is considered as a competing event.
Overall survival (OS) | 54 weeks
  Overall survival is defined as the period from the induction registration to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.
Quality of life during trial | 54 weeks
  Quality of life will be measured by the FACT Lym before start of treatment and during trial participation.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Buske, Prof. Dr., Principal Investigator — University Hospital of Ulm Department of Internal Medicine III
Locations (12):
- Germany (12):
  - Universitätsklinikum Ulm; Klinik für Innere Medizin Innere Medizin III, Ulm, Baden-Wurttemberg
  - Charité Universitätsmedizin Berlin; Hämatologie - Onkologie - Tumorimmunologie, Berlin
  - Klinikum Chemnitz gGmbH, Klinik für Innere Medizin III, Chemnitz
  - Gemeinschaftspraxis Dr. med. Johannes Mohm, Dr. med. Gabriele Prange-Krex, Dresden
  - Kliniken Maria Hilf GmbH; Klinik für Hämatologie, Onkologie und Gastroenterologie, Mönchengladbach
  - Klinikum rechts der Isar der TU München, Klinik und Poliklinik für Innere Medizin III, München
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Klinikum Oldenburg AöR, Universitätsklinik für Innere Medizin, Onkologie und Hämatologie, Oldenburg
  - Brüderkrankenhaus St. Josef, Klinik für Hämatologie und Onkologie, Paderborn
  - Klinikum Passau, II. Medizinische Klinik - Hämatologie, Onkologie und Palliativmedizin, Passau
  - RoMed Klinikum Rosenheim, Med. Klinik II / OTK, Rosenheim
  - Robert-Bosch-Krankenhaus; Hämatologie, Onkologie und Palliativmedizin, Stuttgart